CLINICAL TRIAL: NCT07168057
Title: Young Children and Screens: A Study Protocol of Parents' Perspectives and Child Health Nurses' Approaches in a Digital Age
Brief Title: Young Children and Screens: Parents' Perspectives and Child Health Nurses' Approaches in a Digital Age
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kirsi Tiitinen Mekhail, Pricipal Investigator, Karolinska Institutet
Other Study IDs: Karolinska Inst 2025-03424-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Health Care Providers; Early Childhood Behavior; Child Health Services; Parenting Practices; Caregivers; Nursing Practice
Keywords: digital advisory services; child healthcare; nurses; parents; screen use
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of the research project is to investigate screen habits among children (0-5 years) and their parents including nurses' perspective, and further parents' and nurses' experiences of using web-based healthcare advisory services within Swedish child health care (CHC).

The main research questions are:

What is the correlation between children's and their parents' screen use?

How does screen use differ among families with various socioeconomic backgrounds?

How well does the modified SCREEN-Q instrument measure screen use in Swedish conditions?

How do parents perceive their own and their children's screen use and their parental role?

What are parents' views on available advice and recommendations regarding children's screen use?

How do parents use and experience web-based advisory services within health care and Swedish child health care (CHC)?

How do CHC nurses address screen media-related issues within CHC?

What are CHC nurses' experiences with web-based advisory services?

Participants will:

* Complete a survey on screen habits and digital health service use (N ≈ 300)
* Contribute to validation of a modified SCREEN-Q instrument
* Take part in interviews (parents) and focus groups (child health nurses)

DETAILED DESCRIPTION:
This study investigates screen habits among children aged 0-5 years and their parents, as well as child health nurses' experiences with screen-related guidance and digital health advisory services within Swedish Child Health Care (CHC). The study is grounded in the WHO framework on social determinants of health (1), recognizing that screen use is influenced by individual, familial, and societal factors.

Study Design and Methodology:

A mixed-methods design is employed. The quantitative component consists of a cross-sectional survey (N=300) using a modified version of the SCREEN-Q instrument (2), adapted for Swedish conditions. Psychometric validation will include translation/back-translation, expert review, pilot testing, factor analysis, and reliability testing (Cronbach's alpha). Data will be collected digitally and via paper forms through local Child Health Care centers across three regions in Sweden.

The qualitative component includes two semi-structured interview studies with parents (N=10-15 per sub-study) and focus group discussions with child health nurses (N=15-24 total). These will explore attitudes toward screen use, perceptions of parental roles, and experiences with digital health services. Interviews and discussions will be recorded and transcribed for analysis.

Data Management and Quality Assurance:

All survey data will be stored in REDCap at Karolinska Institutet, locked by passwords. Paper surveys will be stored in locked cabinets. Data validation procedures include automated range and consistency checks. Manual review will be performed for flagged entries. A data dictionary will be developed for all variables, including coding schemes and definitions.

Source data verification will be conducted by comparing survey responses with recruitment logs and consent forms. No external medical records will be used.

Within the project there will be step-by-step procedures to guide how participants are recruited, how informed consent is collected, and how data is gathered, entered, and analyzed. These procedures will also include instructions for handling any unexpected changes in the study or any other issues that may arise.

Sample Size and Statistical Analysis:

A sample size of 300 was determined based on a medium effect size (Cohen's d = 0.5), α = 0.05, and power = 80% (3), sufficient for psychometric validation and subgroup analyses.

Quantitative data will be analyzed using SPSS. Analyses include descriptive statistics, t-tests, ANOVA, chi-square tests, and regression analyses to examine relationships between screen use and background variables. Psychometric validation will include exploratory factor analysis and reliability testing.

Qualitative data will be analyzed using Thematic/content analyses to identify themes and patterns related to screen use and digital health service experiences.

Missing Data Plan:

Missing data will be handled using multiple imputation techniques for quantitative analysis. For qualitative data, incomplete transcripts will be excluded from thematic coding. All procedures will follow ethical guidelines and data protection regulations.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose child/children is/are registered in the Swedish Child Health Care center(s) that participate in the study and that have at least one child at age 0-5 yrs.
* Child health nurses working in the Swedish Child Health Care center(s) that participate in the study

Exclusion Criteria:

* Parent not having children registered in the participating health care centers at age 0-5 yrs.
* Child health nurses not working at the participating child health centers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the cross-sectional (qualitative part of the project) consists of:
  -Parents or primary caregivers of children aged 0-5 years who are enrolled in Child Health Services in Sweden. Participants will be recruited from child health service units located in at least three different regions, including both urban and rural areas, to ensure diversity in geographic and socioeconomic backgrounds.
  Later part of the project includes parents for the same population for qulitative studies. Nurses working in these regions will also be included in the qualitative part of the study to provide professional perspectives on screen use and digital health services.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Parents' screen use | Day 1
  Parents are asked about following in SCREEN-Q (modified):
  Primary place of work or study, Time spent on screen-based work tasks at home on weekdays and weekends, Time spent on screen-based leisure activities on weekdays and weekends, Types of screen-based leisure activities,
Child's screen use | Day 1
  Parents are asked about following in SCREEN-Q (modified):
  Child's Access to Screens, Child's Use of Screen Devices, Child's Ownership of Screen Devices, Time Spent on Screen-Based Activities, Screen Media Habits at Home, Rules for Screen Use, Screen Use During the Day, Multitasking and Social Context of Screen Use, Parental Perceptions of Child's Screen Use, Age When Child Received Own Devices

OTHER OUTCOMES:
Demographic background factors: quantitative study about screens | Day 1
  Parents are asked:
  Age, Gender, Number of children, Age of the child, Family situation, Educational background, Country of birth, Time living in Sweden, Employment status, Relationship to the child, Number of people in the household
Themes identified through semi-structured interviews on parental reasoning and attitudes about screen use | Day 1
  This outcome will be assessed using semi-structured interviews with parents. Interviews will be transcribed and analyzed using thematic analysis or content analyses. The analysis will explore parental motivations, beliefs, and contextual factors influencing screen use. Findings will be reported as descriptive thematic categories.
  Unit of Measure Emergent qualitative themes/categories
Themes identified through interviews on parental perceptions of screen-related guidance and recommendations | Day 1
  This outcome will be assessed through semi-structured interviews with parents, focusing on their perceptions of professional guidance and recommendations regarding children's screen use. Transcripts of audio-recorded interviews will be analyzed using thematic/content analysis to identify key themes such as clarity, usefulness, and trust in guidance received.
  Unit of Measure: Emergent qualitative themes/categories
Demographic background factors for qualitative interviews about digital advisory services | Day 1
  Demographic background factor are asked at the time of interview :
  Parents: Age, Gender, Number of children, Age of the child, Family situation, Educational background, Country of birth, Time living in Sweden, Employment status, Relationship to the child
Themes identified through interviews on parents' experiences with web-based advisory services | Day 1
  Semi-structured interviews will be conducted with parents to explore their experiences using digital advisory services related to screen use. The audio-recorded interviews will be transcribed and analyzed using thematic analysis or content analyses to identify themes/categories related to accessibility, relevance, satisfaction, and barriers to use.
  Unit of Measure: Emergent qualitative themes/categories
Demographic background for focus group discussions with nurses | Day 1
  Nurses: Age, Gender, Region of Employment, Years of Experience as a child health nurse, employment Percentage in Child Health Services, Specialist Education
Short questionnaire about nurses' working methods before focus group discussions | Day 1
  Following areas are covered in the short questionnaire:
  Focus areas, Guidelines used, Knowledge level, Confidence level, Training received, Discussion challenges, Support needs, Regional policies, Training frequency, Experience impact, Trust influence, Web advisory use
Themes identified through focus group discussions with nurses regarding current screen use of families | Day 1
  This outcome will be assessed through focus group discussions with nurses. Discussions will be audio-recorded and thematic analysis/content analyses will be used to identify themes/categories related to current practices, challenges, and strategies in advising families about screen use.
  Unit of Measure: Emergent qualitative themes/categories.

CONTACTS AND LOCATIONS:
Overall Officials: Lise-Lott Rydström, RN., PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared for this study/project. The data include sensitive information about young children and their families, and despite anonymization, there remains a risk of re-identification, particularly in small or region-specific samples. Furthermore, the informed consent obtained from participants does not include provisions for broad data sharing, and ethical approval for such sharing has not been granted.

REFERENCES:
- [Background] 3. Cohen J. Statistical Power Analysis. Current Directions in Psychological Science. 1992;1(3):98-101.
- [Background] Klakk H, Wester CT, Olesen LG, Rasmussen MG, Kristensen PL, Pedersen J, Grontved A. The development of a questionnaire to assess leisure time screen-based media use and its proximal correlates in children (SCREENS-Q). BMC Public Health. 2020 May 12;20(1):664. doi: 10.1186/s12889-020-08810-6. PMID 32397984
- [Background] 1. World Health Organization. (2025). World report on social determinants of health equity. WHO. https://www.who.int/teams/social-determinants-of-health/equity-and-health/world-report-on-social-determinants-of-health-equity
- [Background] Mekhail KT, Blom L, Rydstrom LL. Young children's screen habits and first-time parents' reflections on screen use in socioeconomically disadvantaged Swedish settings: a mixed methods study. BMC Public Health. 2024 Jul 29;24(1):2027. doi: 10.1186/s12889-024-19557-9. PMID 39075392